CLINICAL TRIAL: NCT01762527
Title: Adaptive Radiotherapy Using Plan Selection for Bladder Cancer: A Phase II Trial
Brief Title: Adaptive Radiotherapy Using Plan Selection for Bladder Cancer
Acronym: plan selection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUH-KFE-1217; jr.nr. 1-16-02-283-12 (Other Grant/Funding Number: The Danish National Committee on Health Research Ethics)
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2015-12

CONDITIONS: Adverse Effects for Adaptive RT of Bladder Cancer
Keywords: Adaptive radiotherapy; Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Daily adaptation of radiotherapy
Oversight: Data Monitoring Committee: No

ARMS (1):
- ART (Experimental): Online adaptive radiotherapy
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — CTCAE scoring baseline, every 2'nd week during RT, 2 weeks, 3, 12 and 24 month after RT cineMR (time resolved MR) baseline and weekly during RT for intra fractional motion
  Other Names: Online Adaptive RT using plan selection

SUMMARY:
This protocol describes a Phase 2 clinical trial of online adaptive Radiotherapy, using a library of 3 dose plans corresponding to Small, Medium and Large size bladder. The procedure includes 'Common Toxicity Criteria for Adverse Effects'(CTCAE) for registration of adverse effects (baseline, every 2'nd week during RT, 2 weeks, 3, 6, 12 and 24 month after RT) as well as cineMR for intra-fractional motion (baseline and every week during RT). Patients receive standard non-adaptive RT in the first week. Delineations of the bladder on the Cone-Beam scans (CBCT) from first week of treatment are used for planning the Small and Medium size bladder plans. Large size plan are the standard non-adaptive treatment plan used for the first week of treatment. A margin of 5 mm for intra fractional movement is used.

DETAILED DESCRIPTION:
After inclusion patients are asked about their adverse effects by an oncologist using CTCAE (version 4.0) questionnaire. A planning CT-scan is acquired and for the first 10 patients also a MR-scan for intra fractional motion is acquired. The MR sequence is repeated every week during radiotherapy. The first week of treatment a standard non-adaptive IMRT-plan is used and CBCT-scans are acquired before and after treatment. The CBCT-scans are used for delineation of the bladder on the CBCT-scans from the first 4 fractions. The adaptive plans are generated from the union of the first 4 CBCT-bladders and the planning CT bladder (medium size) and the volume contained in at least 2 out of the 5 bladder volumes (small size). Details can be found in the reference list. From the 6'Th fraction the treatment is performed using the most appropriate size of treatment plan. CTCAE is repeated every other week during radiotherapy and 2 weeks, 3, 6, 12 and 24 month after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven bladder cancer
* Age over 18 years
* Urothelial or planocellular carcinoma
* Stage T2 T4A
* Stage N0M0
* Suitable for radiotherapy
* ECOG/WHO performance status 0-2

Exclusion Criteria:

* Suspected or confirmed distant metastases
* Previous surgery in the small pelvis
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Gastro- Intestinal toxicity | Up to 2 years after ART
  Grade 2 or more GI toxicity using CTCAE 4.0 baseline, every 2'nd week during RT, 2 weeks, 3, 12 and 24 month after RT

SECONDARY OUTCOMES:
Intra-fractional changes of bladder shape and size | spring 2013
  CineMR (time resolved MR) is performed pre-treatment and weekly during RT for the first 10 patients
Difference in accumulated dose to normal tissue | autum 2014
  The gain of normal tissue sparring will be calculated using dose accumulation
1 or 2 years disease free survival | 2015
  1 or 2 years disease free survival will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Morten Høyer, MD, Professor, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Department of Oncology, Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

REFERENCES:
- [Background] Vestergaard A, Sondergaard J, Petersen JB, Hoyer M, Muren LP. A comparison of three different adaptive strategies in image-guided radiotherapy of bladder cancer. Acta Oncol. 2010 Oct;49(7):1069-76. doi: 10.3109/0284186X.2010.501813. PMID 20831498
- [Background] Vestergaard A, Hafeez S, Muren LP, Nill S, Hoyer M, Hansen VN, Gronborg C, Pedersen EM, Petersen JB, Huddart R, Oelfke U. The potential of MRI-guided online adaptive re-optimisation in radiotherapy of urinary bladder cancer. Radiother Oncol. 2016 Jan;118(1):154-9. doi: 10.1016/j.radonc.2015.11.003. Epub 2015 Nov 26. PMID 26631646
- [Result] Vestergaard A, Muren LP, Lindberg H, Jakobsen KL, Petersen JB, Elstrom UV, Agerbaek M, Hoyer M. Normal tissue sparing in a phase II trial on daily adaptive plan selection in radiotherapy for urinary bladder cancer. Acta Oncol. 2014 Aug;53(8):997-1004. doi: 10.3109/0284186X.2014.928419. Epub 2014 Jun 24. PMID 24957559
- [Result] Gronborg C, Vestergaard A, Hoyer M, Sohn M, Pedersen EM, Petersen JB, Agerbaek M, Muren LP. Intra-fractional bladder motion and margins in adaptive radiotherapy for urinary bladder cancer. Acta Oncol. 2015;54(9):1461-6. doi: 10.3109/0284186X.2015.1062138. Epub 2015 Aug 27. PMID 26313410